CLINICAL TRIAL: NCT06973642
Title: Evaluation of Home-based Telerehabilitation Platform to Augment Orthopedic Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Jacob B. Daniels DPT, EdD, Assistant Professor, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UMMC-IRB-2024-178; 6 U66RH31459-06-01 (Other Grant/Funding Number: Department of Health and Human Services: Health Resources and Services Administration)
Record Dates: First submitted 2025-04-11; First posted 2025-05-15 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-04

CONDITIONS: Anterior Cruciate Ligament Reconstruction Rehabilitation
Keywords: telerehabilitation; telehealth; physical therapy; Anterior Cruciate Ligament Rehabilitation

STUDY DESIGN:
Intervention Model Description: Feasibility Criteria
  1. ≥80% of participants will have initial physical therapy visit scheduled within 1 week of enrollment
  2. ≥80% of participants will complete their first physical therapy appointment within 1 week of surgery
  3. Zero major adverse events will result from telehealth physical therapy services
  4. Patient's will complete ≥70% of scheduled physical therapy visits
  5. ≥70% of participants will report satisfaction with telehealth services
  6. >90% of providers will report satisfaction with use of the application to provide rehabilitation services
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation (Experimental): Patient participants will receive telehealth rehabilitation services Provider participants will be providing the physical therapy services.
  Interventions: Device: Software as a Medical Device (WizeCare)

INTERVENTIONS:
Device: Software as a Medical Device (WizeCare) — Telehealth services will be provided through a telerehabilitation platform with AI capabilities and markerless motion capture.

SUMMARY:
The goal of this study is to assess the feasibility of utilizing a telehealth rehabilitation platform to increase patient access for individuals who have undergone orthopedic surgery.

Patient participants will be seen via telehealth until they are able to be seen by an in-person physical therapist of their choice.

Provider participants will be the physical therapist who are providing physical therapy services through the telehealth application.

Data collection:

Patient and provider post surveys Home program and scheduled visit compliance rate Healthcare information in keeping with Stand of care physical therapy practices

Feasibility criteria will be assessed to determine whether this modality improves physical therapy access for patients living in rural areas.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are candidates for anterior cruciate ligament reconstruction.

Exclusion Criteria:

* Visual impairment greater than 20/200 with the use of corrective lenses
* Does not own or have consistent access to a phone with data capabilities
* Has been informed by their healthcare provider that they should not participate in physical therapy services
* Participants can be excluded from the study at any time if the physical therapist determines the patient is not an appropriate candidate for telehealth therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to initial physical therapy visit | At study completion, average 1 year
  Number of days from the time the patient is enrolled in the study until the time they have their first physical therapy visit
Time to first physical therapy visit scheduled | At study completion, average 1 year
  Number of days from when the patient is enrolled to when their first physical therapy visit is scheduled
Number of major adverse events reported from telehealth physical therapy services | Through study completion, an average of 1 year
  Numerical count of how many major adverse events patients or providers report
Number of Scheduled physical therapy visits completed by enrolled patients | At study completion, average 1 year
  Number of scheduled physical therapy sessions completed by patients compared to number of sessions scheduled
Number of participants' surveys that report satisfaction with telehealth services | At study completion, average 1 year
  Participants will complete surveys after each telehealth session. Number of participants' surveys that report satisfaction compared to dissatisfaction will be measured.
Number of providers' surveys that report satisfaction with telehealth application use | At study completion, average 1 year
  Providers will complete surveys after each telehealth session. Number of providers' surveys that report satisfaction compared to dissatisfaction will be measured.

SECONDARY OUTCOMES:
Lower Extremity Functional Scale | Through study completion, an average of 1 year
  Lower Extremity Functional scale is a questionniare designed to assess functional status in patients with Lower extremity problems. The scale is 0-80 with a higher score demonstrating higher functional status
Operative lower extremity pain | Through study completion, an average of 1 year
  Pain in relation to the lower extremity that has undergone ACL reconstructive surgery will be measured on a 0-10 scale with 0 being no pain and 10 being worse pain.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Undecided